CLINICAL TRIAL: NCT06464861
Title: Sequential Treatment With 7x19 CAR-T After Umbilical Cord Blood Derived CD19 CARNK in Relapsed/Refractory B Cell Lymphoma
Brief Title: Sequential Treatment of CD19 CARNK and 7x19 CAR-T in R/R B Cell Lymphoma
Acronym: CD19-CARNK/T
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024 (0673)
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-06

CONDITIONS: Primary Mediastinal B-cell Lymphoma (PMBCL); Mantle Cell Lymphoma (MCL); Diffuse Large B Cell Lymphoma( DLBCL)
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-CAR-NK/T (Experimental): All subjects were intravenously administrated with CAR-NK019 at day 0 with a dose of 2x10^6/kg, and after 1 week will be infused with 7x19 CAR-T at the dose of 2x10^6/kg
  Interventions: Biological: CD19-CAR-NK/T

INTERVENTIONS:
Biological: CD19-CAR-NK/T — Cord blood derived CD19 CARNK sequential Treatment with 7x19 CAR-T

SUMMARY:
To study the safety and efficacy of cord blood-derived CD19 CAR-NK cells sequential with 7x19 CAR-T in relapse / refractory B cell lymphoma

DETAILED DESCRIPTION:
This is a single-center, open, single-arm clinical exploratory study to observe the safety and efficacy of cord blood derived CD19 CAR-NK cells sequential treatment with 7x19 CAR-T in relapse / refractory B cell lymphoma. This study consisted of two phases: phase I: CARNK cells preparation and infusion (Day0, dose of 2 x 10^6 / kg). Phase II: 7x19 CAR-T cells preparation and infusion (Day7, dose 2×10^6/kg).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, no gender limit;
2. Histologically diagnosed as diffuse large B-cell lymphoma (DLBCL), transforming follicular lymphoma (TFL), primary mediastinal B-cell lymphoma (PMBCL), mantle cell lymphoma (MCL) and other inert B-cells NHL conversion type:

   1. Refractory or relapsed DLBCL refers to the failure to achieve complete remission after 2-line treatment; disease progression during any treatment, or disease stable time equal to or less than 6 months; or disease progression or recurrence within 12 months after autologous hematopoietic stem cell transplantation ；
   2. Refractory or relapsed MCL must be resistant to or intolerable to BTK inhibitors;
   3. Refractory or relapsed indolent B-cell NHL is the failure or recurrence of third-line treatment;
3. Previous treatment must include CD20 monoclonal antibody treatment (unless the subject is CD20 negative) and anthracyclines;
4. At least one measurable lesion with the longest diameter ≥ 1.5 cm exists;
5. The expected survival period is ≥12 weeks;
6. The puncture section of the tumor tissue was positive for CD19 expression;
7. ECOG score 0-2 points;
8. Sufficient organ function reserve:

   1. Alanine aminotransferase, aspartate aminotransferase ≤ 2.5× UNL (upper limit of normal value);
   2. Creatinine clearance rate (Cockcroft-Gault method) ≥60 mL/min;
   3. Serum total bilirubin and alkaline phosphatase ≤1.5× UNL;
   4. Glomerular filtration rate>50Ml/min
   5. Cardiac ejection fraction (EF) ≥50%;
   6. Under natural indoor air environment, basic oxygen saturation>92%
9. Allow a previous stem cell transplantation
10. The approved anti-B-cell lymphoma treatments, such as systemic chemotherapy, systemic radiotherapy, and immunotherapy, have been completed for at least 3 weeks before the study medication;
11. Allow patients who have previously received CAR-T cell therapy and have failed or relapsed after 3 months of evaluation;
12. Female subjects of childbearing age must have a negative pregnancy test and agree to take effective contraceptive measures during the trial
13. Two tests for the new coronavirus or swine flu virus are negative.

Exclusion Criteria:

1. Allergic to any of the components of cell products;
2. History of other tumors;
3. Acute GvHD or extensive chronic GvHD with grade II-IV (Glucksberg standard) in the past or are receiving anti-GVHD treatment;
4. Had received gene therapy within the past 3 months;
5. Active infections requiring treatment (except for simple urinary tract infections, bacterial pharyngitis); however, prophylactic antibiotics, antiviral and antifungal infection treatment are permitted;
6. Patents infected with hepatitis B (HBsAg positive, but HBV-DNA < 103 is not excluded) or hepatitis C virus (including virus carriers), syphilis and other acquired and congenital immunodeficiency diseases, including but not limited to HIV-infected persons;
7. Subjects with Grade III or IV cardiac dysfunction according to the New York Heart Association's cardiac function grading criteria;
8. Patients who received antitumor therapy earlier but did not recover from the toxicity (CTCAE 5.0 toxicity did not recover to ≤ grade 1, except fatigue, anorexia, alopecia);
9. Subjects with a history of epilepsy or other central nervous system disorders;
10. Head-enhanced CT or MRI showing evidence of central nervous system lymphoma;
11. Lactating women who are unwilling to stop breastfeeding;
12. Any other factors that the investigator believes may increase the risk to the subject or interfere with the test results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | Up to 28 days
  To evaluate the safety and tolerability of cord blood-derived anti-CD19 CAR-NK Cell sequential with 7X19 CAR-T for B-cell Non-Hodgkin Lymphoma

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 2 years
  To determine the OS of CB CD19 CAR-NK Cell sequential with 7X19 CAR-T for B-cell Non-Hodgkin Lymphoma
Progression free survival (PFS) | Up to 2 years
  To determine the anti-tumor efficacy of CB CD19 CAR-NK Cell sequential with 7X19 CAR-T for B-cell Non-Hodgkin Lymphoma
Duration of response (DOR) | Up to 2 years
  To determine the DOR of CB CD19 CAR-NK Cell sequential with 7X19 CAR-T for B-cell Non-Hodgkin Lymphoma
Complete response rate (CR) | Up to 2 years
  To determine the CR rate of CB CD19 CAR-NK Cell sequential with 7X19 CAR-T for B-cell Non-Hodgkin Lymphoma
Partial response rate (PR) | Up to 2 years
  To determine the PR rate of CB CD19 CAR-NK Cell sequential with 7X19 CAR-T for B-cell Non-Hodgkin Lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Wenbin, Professor, Study Chair — Zhejiang University
Locations (1):
- the Second Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No